CLINICAL TRIAL: NCT05509855
Title: A Long-Term Safety Follow-Up Study for Patients Treated With Anti-CD7 Allogeneic CAR-T Cells (WU-CART-007)
Brief Title: A Long-Term Safety Follow-Up Study for Patients Treat With WU-CART-007
Status: Enrolling by invitation | Type: Observational
Sponsor: Wugen, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: WUC007-02
Record Dates: First submitted 2022-07-20; First posted 2022-08-22 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; T-cell Lymphoblastic Lymphoma
Keywords: T-ALL; T-LBL
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Test for replication-competent lentivirus (RCL) and cellular persistence following treatment with WU-CART-007 will be performed until cells are undetectable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with WU-CART-007: Patients who received previous treatment with WU-CART-007
  Interventions: Genetic: Genetic: WU-CART-007

INTERVENTIONS:
Genetic: Genetic: WU-CART-007 — No study drug is administered in this study. Patients who have received WU-CART-007 will be enrolled in this study for Long Term Safety and Efficacy

SUMMARY:
This study will provide long-term follow-up for patients who have received treatment with WU-CART-007 in a previous clinical trial. In this study, patients will be followed for up to 15 years after their last dose of WU-CART-007 for evaluation of delayed adverse events, presence of persisting WU-CART-007 vector sequences, and overall survival and progression-free survival.

DETAILED DESCRIPTION:
This long-term follow-up (LTFU) study is designed to follow patients for up to 15 years after WU-CART-007 infusion to evaluate the persistence of the WU-CART-007 cell clones and to explore any unanticipated genetic consequences secondary to the introduction of genetically modified cells. Long-term toxicity, subsequent anti-cancer therapy, and survival status will be monitored.

Patients will transition to this LTFU study when they meet the criteria for discontinuation from the main study or after completing 24 months of follow-up in the main study. Patients will be contacted every 6 months for the first 5 years following WU-CART-007 administration and then yearly, for up to 10 years, for a total of 15 years of follow-up after prior WU-CART-007 treatment or until death, whichever occurs first.

Patients will be evaluated either at the treating site or by the patient's primary Health Care Provider (HCP). Patients will be required to allow key sponsor contacts to continue to access medical records so that information related to their health condition and initial treatment response may be obtained.

ELIGIBILITY:
Inclusion Criteria: Patients that received WU-CART-007 in the context of any investigational study will be eligible to participate in this long-term follow-up study.

Exclusion Criteria: Not Applicable

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient population will consist of patients who participated in a previous clinical trial where WU-CART-007 was administered.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2037-07-01 (Estimated); Study Completion 2037-07-01 (Estimated)

PRIMARY OUTCOMES:
Delayed adverse events (AEs)/serious adverse events (SAEs) | up to 15 years
  assess the risk of delayed adverse events including serious events following exposure to WU-CART-007
Persistence of WU-CART-007 cells | Every 6 months for up to 5 years and then yearly for up to 15 years
  Peripheral blood samples will be monitored used polymerase chain reaction for persistence of WU-CART-007 cells
Tanner Staging | up to 15 years
  Tanner Staging will be used to evaluate growth and development outcomes and sexual maturity status for patients who were < 18 years of age at the time of treatment with WU CART-007

SECONDARY OUTCOMES:
Overall survival (OS) | up to 15 years
  To evaluate survival n patients previously treated with WU-CART-007
Progression-free survival (PFS) | up to 15 years
  To evaluate profession free survival in patients previously treated with WU-CART-007

CONTACTS AND LOCATIONS:
Overall Officials: Cherry Thomas, MD, Study Director — Wugen, Inc.
Locations (5):
- United States (4):
  - City of Hope, Duarte, California
  - Childrens Hospital LA, Los Angeles, California
  - Washington University, St Louis, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Peter MacCullam Cancer Center, Melbourne, Australia